CLINICAL TRIAL: NCT06795100
Title: Pharmacokinetic Study of Intravenous Lidocaine in Young and Elderly Patients
Acronym: ElderLIDO_1
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC23_9774_07_ElderLIDO_1
Record Dates: First submitted 2024-12-13; First posted 2025-01-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elderly patients (Other): Adult participant ≥ 70 years old
  Interventions: Other: Pre-inclusion; Other: Inclusion; Drug: Lidocaine; Other: Pharmacokinetic study of intravenous lidocaine; Other: Pain; Other: adverse effects/events; Biological: biological blood test
- Young patients (Other): Adult participant ≤ 40 years old)
  Interventions: Other: Pre-inclusion; Other: Inclusion; Drug: Lidocaine; Other: Pharmacokinetic study of intravenous lidocaine; Other: Pain; Other: adverse effects/events; Biological: biological blood test

INTERVENTIONS:
Other: Pre-inclusion — Information and presentation of the proposed study to participants during the anesthesia consultation scheduled prior to surgery, including provision of the information document and consent form. Trial participants will have at least 2 days to decide whether or not to take part in the trial.
Other: Inclusion — Participants will be welcomed according to the usual process in the digestive, hepatic, urological, or gynecological surgery service. The inclusion visit will coincide with the pre-anesthesia visit during which the absence of contraindications for starting the study will be verified, particularly the occurrence of any health changes since the anesthesia visit that would contraindicate anesthesia or lidocaine administration. During this visit, participant consent will be obtained. The informed consent form must be signed no later than the morning of the intervention.
  For women of childbearing age, the absence of current pregnancy will be verified orally for each participant included. A pregnancy test may be performed if the participant so wishes, but a systematic test is not justified.
Drug: Lidocaine — Induction of anesthesia will be at the discretion of the attending anesthesiologist, with a lidocaine bolus of 2 mg/kg administered over 1 minute, followed by a continuous IV infusion of 2 mg/kg/h.
Other: Pharmacokinetic study of intravenous lidocaine — Blood samples of 3 mL will be collected in heparinized tubes without gel of 4 ml at 30, 60 and 120 minutes after the start of lidocaine infusion, then every two hours during surgery, and two finals samples at 15 and 60 minutes after the infusion stops.
Other: Pain — . Maximal pain reported in the post-anesthesia care unit (PACU) and maximal pain at rest and with movement at 24 hours post-extubation will be recorded.
Other: adverse effects/events — Any adverse effects/events will be documented from the start of lidocaine administration until 24 hours post-extubation,
Biological: biological blood test — A biological blood test, not performed in routine practice, will be carried out to measure the following parameters: albumin, ASAT, ALAT, PAL, GammaGT, total and conjugated bilirubin, creatinine, with calculation of GFR.

SUMMARY:
Aging is accompanied by a gradual alteration in the functional reserve of several organs and a change in body composition that can affect the pharmacokinetics, response, and safety profile of medications. Lidocaine is a local anesthetic used daily in perineural or intravenous administration to reduce the need for opioids. Although its analgesic efficacy is well-established, there is currently only one older study regarding the pharmacokinetics and pharmacokinetic-pharmacodynamic (PK-PD) relationship of lidocaine in healthy elderly patients. In this study, conducted with a small sample size (13 subjects over 64 years old and 24 young subjects under 38 years old) and using a low bolus of 25 mg, the half-life of lidocaine was increased by 59% and clearance was decreased by 35% in elderly male subjects without significant differences in females. However, the recommendations for intravenous administration of lidocaine for analgesic purposes are the same for all: a bolus of 1 to 2 mg/kg followed by continuous administration of 1.5 to 2 mg/kg/h. Morphine sparing is particularly important in elderly patients due to their increased sensitivity to adverse effects. With this study, the investigators aim to define the optimal dose to administer in elderly subjects, in order to optimize analgesia while remaining within the therapeutic range to limit the adverse effects of lidocaine.

ELIGIBILITY:
Inclusion Criteria:

CI1 - Adult participant (≤ 40 years old) and (≥ 70 years old). CI2 - Undergoing abdominal, digestive, hepatic, urological, or gynecological surgery with an expected duration > 2 hours.

CI3 - Covered by a social security plan. CI4 - Provided with both oral and written information about the protocol and has signed informed consent to participate in this research.

Exclusion Criteria:

NC1 - Allergy to lidocaine or any of its excipients.

NC2 - Presence of comorbidities that may alter lidocaine pharmacokinetics, such as:

* Heart failure (ejection fraction < 45%).
* Renal failure (creatinine clearance < 15 ml/min).
* Hepatic failure (prothrombin time < 15%).
* Body Mass Index (BMI) > 30.

NC3 - Long-term treatment with an antiarrhythmic drug.

NC4 - Ongoing treatment with strong CYP 1A2 inhibitors (e.g., Ciprofloxacin, Fluvoxamine) and/or CYP 1A2 inducers (e.g., Carbamazepine, Modafinil, Ritonavir).

NC5 - Use of peripheral or neuraxial regional anesthesia or local anesthetic infiltration.

NC6 - Known pregnancy or ongoing breastfeeding.

NC7 - Adult under legal protection (e.g., judicial safeguard, guardianship, or tutelage) or deprived of liberty.

NC8 - Participation in another interventional study.

EXCLUSION CRITERIA

EC1 - Any eligibility criterion that is no longer met between the signing of consent and the day of surgery.

EC2 - Participant with no blood sample for pharmacokinetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of lidocaine | at 60 min from initial lidocaine bolus
  Plasma concentration of lidocaine at steady state ( at 60 min from initial lidocaine bolus)

SECONDARY OUTCOMES:
Clearance | Day 0
  Other pharmacokinetic parameters of lidocaine: clearance
Area under the curve | Day 0
  Other pharmacokinetic parameters of lidocaine: area under the curve (AUC)
plasma half-life | Day 0
  Other pharmacokinetic parameters of lidocaine: plasma half-life
Volume of distribution | Day 0
  Other pharmacokinetic parameters of lidocaine: volume of distribution.
Free concentration | Day 0
  Free concentration of lidocaine.
Total morphine-equivalent consumption | 24 hours post-extubation.
  Total morphine-equivalent consumption at 24 hours post-extubation.
Maximal pain reported in the post-anesthesia care unit (PACU) | Day 0
  Maximal pain reported in the post-anesthesia care unit (PACU) assessed using the Numerical Rating Scale (NRS) for pain (Numerical scale from 0 to 10 (0: no pain, 10: worst pain ever experienced))
Maximal pain at rest in the 24h post-extubation | 24 hours post-extubation
  Maximal pain at rest in the 24h post-extubation, assessed using the Numerical Rating Scale (NRS) for pain. (Numerical scale from 0 to 10 (0: no pain, 10: worst pain ever experienced))
Maximal pain with movement in the 24h post-extubation | 24 hours post-extubation
  Maximal pain with movement in the 24h post-extubation, assessed using the Numerical Rating Scale (NRS) for pain (Numerical scale from 0 to 10 (0: no pain, 10: worst pain ever experienced))
Frequency of adverse effects | 24 hours post-extubation
  Frequency of adverse effects attributable to lidocaine at 24 hours post-extubation.
Number of adverse effects | 24 hours post-extubation
  Number of adverse effects attributable to lidocaine at 24 hours post-extubation.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, CHU de Rennes
  - CHU de Rennes - Hôpital Sud, Rennes

IPD SHARING:
Plan to Share IPD: Undecided